CLINICAL TRIAL: NCT01741376
Title: Progesterone and Atomoxetine for Cocaine Cessation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: All clinical trials within the Department of Psychiatry at UMN were suspended and this study was withdrawn due to no enrollment.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1P50DA033942-01 (NIH)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Cocaine Dependence; Nicotine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Tobacco Use Disorder | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo + Placebo (Placebo Comparator): Two placebos are given for 84 days.
  Interventions: Drug: Placebo
- Progesterone + Placebo (Active Comparator): Progesterone (200 mg twice daily) and a placebo are given
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Progesterone 200 mg twice daily
  Arms: Progesterone + Placebo
Drug: Placebo
  Arms: Placebo + Placebo

SUMMARY:
The purpose of this study is to examine the role of progesterone (a hormone found in both men and women) on stopping cocaine use. The study will examine whether the medication, in combination with behavior therapy will decrease cocaine use, cigarette smoking, withdrawal symptoms, impulsivity and stress.

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 and 45 and males between 18 and 60 years-of-age;
* Understand the study procedures and provide written informed consent;
* Meet DSM-IV criteria for cocaine or methamphetamine and nicotine dependence;
* Minimum of cocaine use 4 days/months over last 3 months;
* Minimum of 5 cigarettes/day for last twelve months;
* Stable psychiatric status;
* Stable medical status; Willing to use double-barrier contraception method if sexually active and not surgically sterilized;
* Regular menstrual cycles (for females);
* No contraindications to progesterone treatment;
* Ability to participate fully in research elements for the duration of the trial.

Exclusion Criteria:

* DSM-IV diagnoses for current or lifetime psychotic disorders (unless substance induced), bipolar disorder, current ADHD and other current substance dependence (except nicotine dependence, or alcohol or cannabis dependence not exhibiting withdrawal or other features requiring medical attention);
* Currently using nicotine pharmacotherapy preparations;
* history of thromboembolic events, diabetes, stroke, heart disease;
* Psychotropic medications other than stable doses of anti-depressants;
* Currently pregnant or nursing;
* Liver enzyme levels three times normal limits;
* Previous treatment with or adverse response to progesterone.
* Serious suicide attempt within preceding 2 years;
* Current use of exogenous hormones.
* Conditions contraindicated to progesterone treatment (including, but not limited to, thrombophlebitis, deep vein thrombosis, pulmonary embolus, clotting or bleeding disorders, heart disease, diabetes, history of stroke, allergy to peanuts, hypersensitive to progesterone and liver dysfunction).
* History of pheochromotytoma or narrow angle glaucoma,
* Current hypertension, tachycardia or clinically relevant ECG abnormalites;
* Allergy to peanuts,
* Current suicidality or need for emergency psychiatric treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cocaine Cessation | Days 1 to 86
  Urine Test

SECONDARY OUTCOMES:
Impulsivity | Days 1 to 86
  Self report of the following subjective questionnaires: (1) Behavioral Inhibition Activation Scales, (2) Barratt Impulsivity Scale, and (3) Brief Self Control Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M Specker, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No